CLINICAL TRIAL: NCT06252025
Title: The Effect of an Immersive VR Reminiscence System for Facilitating Memory Retrieval Among Nursing Home Older Adults
Brief Title: Immersive VR Reminiscence System for Facilitating Memory Retrieval Among Nursing Home Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhu Dian (Other)
Responsible Party: Sponsor-Investigator, Zhu Dian, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Sjtu0003
Record Dates: First submitted 2024-01-24; First posted 2024-02-09 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Memory, Repressed; Emotional Regulation; Old Age
Keywords: Virtual Reality; Reminiscence Therapy
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR reminiscence therapy system "Memo-gration" (Experimental): This study tailored a variety of instructional material within each virtual scenario, taking into account various memory triggers. Guidance is activated when the user is identified as making physical contact with an object or discussing a specific keyword. This encompasses textual assistance provided within the virtual environment, the display of multimedia information, and the provision of organized voice guidance. Following the system's instructions, users engaged in discussion with the caregiver, and had the freedom to terminate the conversation at their discretion and explore other topics by interacting with different items.
  Interventions: Combination Product: Memo-gration
- Picture reminiscence therapy (Active Comparator): The picture reminiscence therapy group utilized a series of color images depicting screenshots of the Memo-gration, ensuring that the screenshots remained as consistent as feasible with the presented memory cues.
  Interventions: Other: Picture reminiscence therapy

INTERVENTIONS:
Combination Product: Memo-gration — This study tailored a variety of instructional material within each virtual scenario, taking into account various memory triggers. Guidance is activated when the user is identified as making physical contact with an object or discussing a specific keyword. This encompasses textual assistance provided within the virtual environment, the display of multimedia information, and the provision of organized voice guidance. Following the system's instructions, users engaged in discussion with the caregiver, and had the freedom to terminate the conversation at their discretion and explore other topics by interacting with different items.
  Arms: VR reminiscence therapy system "Memo-gration"
Other: Picture reminiscence therapy — Picture reminiscence therapy
  Arms: Picture reminiscence therapy

SUMMARY:
A VR game "Memo-gration" was designed to assist elderly people in reminiscence therapy. The ultimate scene design was crafted in a vintage Chinese aesthetic reminiscent of the previous century.

DETAILED DESCRIPTION:
This study tailored a variety of instructional material within each virtual scenario, taking into account various memory triggers. Guidance is activated when the user is identified as making physical contact with an object or discussing a specific keyword. This encompasses textual assistance provided within the virtual environment, the display of multimedia information, and the provision of organized voice guidance. Following the system's instructions, users engaged in discussion with the caregiver, and had the freedom to terminate the conversation at their discretion and explore other topics by interacting with different items.

ELIGIBILITY:
Inclusion Criteria:

* (i) absence of significant cognitive impairment, visual impairment, hearing impairment, and communication ability.
* (ii) Obtained the pre-test and watched the film while wearing a VR headgear without experiencing any notable discomfort.

Exclusion Criteria:

* (i) Older adults with cognitive impairments that prevent normal communication
* (ii) Visually impaired

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | baseline and 1 day (study completion)
  POMS is utilized to evaluate alterations in affective state and cognitive state induced by short-term psychotherapy, emotional stimuli, etc.Participants assessed their present mental state using a 5-point Likert scale, comprising 40 questions that encompassed 7 subscales measuring tension, despair, weariness, and self-esteem, etc. A comprehensive mood disturbance score (TMD) was ultimately synthesized.

SECONDARY OUTCOMES:
Questionnaire on VR Experience | 1 day (study completion)
  The UMUX-Lite and Slater-Usoh-Steed Proximity Questionnaires are combined to investigate the user experience of older persons with Memo-gration. Both assessments employ a 7-point Likert scale format.

CONTACTS AND LOCATIONS:
Overall Officials: Dian Zhu, Dr, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Dian Zhu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No